CLINICAL TRIAL: NCT01431144
Title: The Effect of Implant Placement and Simultaneous Soft Tissue Augmentation in the Esthetic Zone Using Either Connective Tissue Autograft or Acellular Dermal Matrix Allograft on Peri-implant Hard and Soft Tissue Healing
Brief Title: Implant Placement With Simultaneous Gum Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Henry Greenwell, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11.0355
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2013-07

CONDITIONS: Edentulous
Keywords: soft tissue thickness; dental implant; soft tissue recession; implant exposure
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connective tissue autograft (Active Comparator): A connective tissue autograft harvested from the palate was grafted onto the facial of a simultaneously placed dental implant and soft tissue thickness was measured at baseline and Time 4.
  Interventions: Procedure: connective tissue autograft
- connective tissue allograft (Experimental): An acellular dermal matrix allograft was grafted on the facial surface of a simultaneously placed dental implant and soft tissue thickness was measured at baseline and Time 4.
  Interventions: Procedure: connective tissue allograft

INTERVENTIONS:
Procedure: connective tissue autograft — A connective tissue autograft is harvested from the palate and grafted at the site of implant placement on the facial surface.
  Arms: Connective tissue autograft
Procedure: connective tissue allograft — An acellular dermal matrix allograft (Alloderm, BioHorizons, Inc, Birmingham, AL, USA) is grafted at the site of implant placement on the facial surface.
  Arms: connective tissue allograft

SUMMARY:
This study is a comparison of implant placed and simultaneously grafted with either autogenous connective tissue or a connective tissue allograft. The objective is to determine the change in soft tissue thickness and determine if a better result is obtained with the autograft or the allograft. The hypothesis is that there will be no difference in soft tissue thickness over the implant between the autograft and the allograft technique.

ELIGIBILITY:
Inclusion Criteria:

* One edentulous site bordered by 2 teeth needing a dental implant

Exclusion Criteria:

* Systemic diseases that affect the periodontium
* Previous head and neck radiation
* Smoking more that 1/2 pack per day
* Requires prophylactic antibiotics
* Allergy to meds used in study
* Previous chemotherapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic, School of Dentistry, University of Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 patients were entered, 13 for the test allograft group and 14 for the positive control connective tissue autograft group
Pre-assignment Details: There were no exclusions prior to assignment or treatment.
Groups:
- Connective Tissue Allograft: A connective tissue allograft was placed simultaneously with dental implant placement and soft tissue thickness was measured at baseline and Time 4.
- Connective Tissue Autograft: A connective tissue autograft was placed simultaneously with dental implant placement and soft tissue thickness was measured at baseline and Time 4.
Period: Overall Study
Arm/Group | Connective Tissue Allograft | Connective Tissue Autograft
Started | 13 | 14
Completed | 11 | 14
Not Completed | 2 | 0
Not completed — Implant mobility and removal | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Connective Tissue Allograft | Connective Tissue Autograft | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (21) | 57 (10) | 52 (16)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Soft Tissue Thickness Over the Implant
Description: Soft tissue thickness at the facial osseous crest.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Connective Tissue Allograft | Connective Tissue Autograft
Number analyzed (Participants) | 11 | 14
mm | 0.6 (1.2) | 0.4 (0.7)

ADVERSE EVENTS:
Time Frame: Baseline to final, no adverse events
Arm/Group | Connective Tissue Allograft | Connective Tissue Autograft
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
There were no adverse events. There were 2 cases of implant mobility and these was treated as a potential expected complication and handled with routine clinical practice guidelines.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No